CLINICAL TRIAL: NCT03252353
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled, Multicenter Study to Evaluate Efficacy and Safety of Octreotide Capsules in Patients Who Demonstrated Biochemical Control on Injectable Somatostatin Receptor Ligands (SRL) Treatment
Brief Title: Efficacy and Safety of Octreotide Capsules (MYCAPSSA) in Acromegaly
Acronym: OPTIMAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Chiasma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OOC-ACM-303
Record Dates: First submitted 2017-08-10; First posted 2017-08-17 (Actual); Results first posted 2020-10-19 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Acromegaly
Keywords: Octreotide Capsules, Acromegaly, OPTIMAL, MYCAPSSA
MeSH Terms: conditions — Acromegaly | interventions — Octreotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Octreotide capsules (Active Comparator): Octreotide capsules
  Interventions: Drug: octreotide capsules
- Matching Placebo (Placebo Comparator): Matching placebo capsules
  Interventions: Drug: Matching placebo

INTERVENTIONS:
Drug: octreotide capsules — octreotide capsules 40 mg/day, 60 mg/day, 80 mg/day (individual dose titration)
  Other Names: MYCAPSSA
  Arms: Octreotide capsules
Drug: Matching placebo — Matching placebo capsules
  Other Names: Placebo
  Arms: Matching Placebo

SUMMARY:
Octreotide capsule is a novel, orally-administered formulation of the commercially-available injectable drug octreotide. In a recent phase 3 trial, oral octreotide capsules demonstrated maintenance of biochemical response up to 13 months in the majority of patients with acromegaly previously managed with somatostatin analog injections (reference below).

DETAILED DESCRIPTION:
This is a double blind, randomized study that assesses the efficacy and safety of octreotide capsules vs. placebo. Eligible acromegaly patients, treated with injectable somatostatin analogs, who are biochemically controlled and have prior evidence of active disease, will be randomized to receive either octreotide capsules or placebo for up to 36 weeks. At the end of this double blind, placebo controlled period, eligible patients will receive octreotide capsules in an open-labeled extension for at least one year. Patients failing to respond (per protocol), to oral treatment, (either placebo or octreotide capsules), will be rescued with the standard of care and upon meeting the eligibility criteria could also enroll into the long term extension with octreotide capsules.

This study received agreement from the FDA, under a special protocol assessment.

ELIGIBILITY:
Inclusion Criteria:

* Documented evidence of active acromegaly
* Treatment with Somatostatin analogs injections (octreotide or lanreotide) for at least 6 months with a stable dose for at least the last three months of therapy
* Biochemically controlled

Exclusion Criteria:

* Patients taking injections of long-acting Somatostatin Receptor Ligands (SRLs) not as indicated in the label
* Pituitary surgery within six months
* Conventional or stereotactic pituitary radiotherapy any time in the past
* Patients who previously participated in CH-ACM-01 or OOC-ACM-302
* Any clinically significant uncontrolled concomitant disease
* Symptomatic cholelithiasis
* Pegvisomant, within 24 weeks
* Dopamine agonists, within 12 weeks
* Pasireotide, within 24 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2019-06-13 (Actual); Study Completion 2022-05 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Susan L Samson, MD PhD, Study Chair — Pituitary Center at Baylor St. Luke's Medical
Locations (60):
- United States (19):
  - Keck Medical Center of University of Southern California, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - Stanford University School of Medicine, Palo Alto, California
  - University of Colorado, Aurora, Colorado
  - The Emory Clinic, Atlanta, Georgia
  - John H. Stroger Jr. Hospital of Cook County, Chicago, Illinois
  - Johns Hopkins University Clinical Trials Unit, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Washington University School of Medicine, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Allegheny Endocrinology Associates, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - Huntsman Cancer Hospital, Salt Lake City, Utah
- Australia (6):
  - St Vincent's Private Hospital-NSW, Darlinghurst, New South Wales
  - Royal North Shore Public Hospital, St Leonards, New South Wales
  - St Vincent's Hospital-VIC, Fitzroy, Victoria
  - The Alfred, Melbourne, Victoria
  - Melbourne Health, Parkville, Victoria
  - Keogh Institute (Sir Charles Gardner), Nedlands, Western Australia
- University Specialized Hospital for Active Treatment of Endocrinology "Acad. Iv. Pencev" EAD, Sofia, Bulgaria
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - St Joseph's Health Care, London, Ontario
  - McGill University Health Centre, Montreal, Quebec
- Denmark (2):
  - Aarhus University Hospital, Aarhus
  - Rigshospitalet The Department of Endocrinology, Copenhagen
- Germany (2):
  - RWTH Aachen University Hospital, Medical Clinic III Division of Endocrinology and Diabetes, Aachen
  - Klinikum der LMU Muenchen, Medizinische Klinik und Poliklinik IV, Endokrinologie, Munich
- Hungary (3):
  - Magyar Honvedseg Egeszsegugyi Kozpont, II. sz. Belgyogyaszati Osztaly, Budapest
  - University of Semmelweiss, Budapest, Budapest
  - Szegedi Tudományegyetem, I. Belgyógyászati Klinika, Szeged
- Israel (3):
  - Hadassah Ein-Karem Medical Center, Jerusalem
  - Rabin Medical Center, Beilinson Hospital, Petah Tikva
  - Tel Aviv Sourasky Medical Center, Tel Aviv
- Italy (2):
  - Policlinico di Monserrato U.O.C. Endocrinologia e Diabetologia, Monserrato
  - Azienda Ospedaliero-Universitaria Pisana, Università di Pisa, Pisa
- Riga Eastern Clinical University, Hospital Gailezers Department of Endocrinology, Riga, Latvia
- Netherlands (2):
  - Leids Universitair Medisch Centrum, Leiden
  - Erasmus Medisch Centrum, Rotterdam
- New Zealand (2):
  - Dunedin Hospital, Dunedin
  - Wellington Hospital, Wellington
- Poland (5):
  - Katedra i Klinika Endokrynologii i Chorob Wewnetrznych, Gdansk
  - Uniwersyteckie Centrum Okulistyki i Onkologii Samodzielny Publiczny Szpital Kliniczny Slaskiego Uniwersytetu Medycznego w Katowicach, Oddzial Endokrynologii, Katowice
  - Szpital Uniwersytecki w Krakowie, Oddzial Kliniczny Endokrynologii, Krakow
  - Klinika Chorob Wewnetrznych i Endokrynologii, Warsaw
  - Samodzielny Publiczny Szpital Kliniczny nr 1 we Wroclawiu, Klinika Endokrynologii, Diabetologii i Leczenia Izotopami, Wroclaw
- Medical University Centre Ljubljana, Ljubljana, Slovenia
- Sahlgrenska University Hospital, Gothenburg, Sweden
- Turkey (Türkiye) (4):
  - Ankara University, Faculty of Medicine, Ankara
  - Hacettepe University Medical School, Ankara
  - Ege University Medical Faculty Internal Diseases, Izmir
  - Erciyes University Medical Faculty, Kayseri
- United Kingdom (3):
  - University Hospitals Birmingham NHS Foundation Trust, Queen Elizabeth Hospital, Birmingham
  - Central Manchester University Hospitals NHS Foundation Trust, Manchester Royal Infirmary, Manchester
  - Royal Victoria Infirmary, Newcastle upon Tyne

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Melmed S, Popovic V, Bidlingmaier M, Mercado M, van der Lely AJ, Biermasz N, Bolanowski M, Coculescu M, Schopohl J, Racz K, Glaser B, Goth M, Greenman Y, Trainer P, Mezosi E, Shimon I, Giustina A, Korbonits M, Bronstein MD, Kleinberg D, Teichman S, Gliko-Kabir I, Mamluk R, Haviv A, Strasburger C. Safety and efficacy of oral octreotide in acromegaly: results of a multicenter phase III trial. J Clin Endocrinol Metab. 2015 Apr;100(4):1699-708. doi: 10.1210/jc.2014-4113. Epub 2015 Feb 9. PMID 25664604
- [Background] Tuvia S, Atsmon J, Teichman SL, Katz S, Salama P, Pelled D, Landau I, Karmeli I, Bidlingmaier M, Strasburger CJ, Kleinberg DL, Melmed S, Mamluk R. Oral octreotide absorption in human subjects: comparable pharmacokinetics to parenteral octreotide and effective growth hormone suppression. J Clin Endocrinol Metab. 2012 Jul;97(7):2362-9. doi: 10.1210/jc.2012-1179. Epub 2012 Apr 26. PMID 22539587
- [Derived] Labadzhyan A, Nachtigall LB, Fleseriu M, Gordon MB, Molitch M, Kennedy L, Samson SL, Greenman Y, Biermasz N, Bolanowski M, Haviv A, Ludlam W, Patou G, Strasburger CJ. Oral octreotide capsules for the treatment of acromegaly: comparison of 2 phase 3 trial results. Pituitary. 2021 Dec;24(6):943-953. doi: 10.1007/s11102-021-01163-2. Epub 2021 Jun 25. PMID 34173129
- [Derived] Samson SL, Nachtigall LB, Fleseriu M, Gordon MB, Bolanowski M, Labadzhyan A, Ur E, Molitch M, Ludlam WH, Patou G, Haviv A, Biermasz N, Giustina A, Trainer PJ, Strasburger CJ, Kennedy L, Melmed S. Maintenance of Acromegaly Control in Patients Switching From Injectable Somatostatin Receptor Ligands to Oral Octreotide. J Clin Endocrinol Metab. 2020 Oct 1;105(10):e3785-97. doi: 10.1210/clinem/dgaa526. PMID 32882036
- See also: Chiasma Web Page — http://www.chiasmapharma.com/
- See also: Melmed et al. JCEM 2015 — https://www.ncbi.nlm.nih.gov/pubmed/25664604

RESULTS

PARTICIPANT FLOW:
Groups:
- Octreotide Capsules: Octreotide capsules
  octreotide capsules: octreotide capsules 40mg/day, 60mg/day, 80 mg/day (individual dose titration)
Period: Overall Study
Arm/Group | Octreotide Capsules | Matching Placebo
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Octreotide Capsules | Matching Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 55.3 (11.97) | 54.2 (10.96) | 54.7 (11.38)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 14 | 30
  Male | 12 | 14 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 3 | 3
  Not Hispanic or Latino | 28 | 25 | 53
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 27 | 24 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Baseline average Insulin-like Growth Factor 1 (IGF-1) (categorical) [Count of Participants; unit: Participants]
  IGF≤ 1 Upper Limit of Normal (ULN) | 27 | 23 | 50
  IGF > 1 to < 1.3 ULN | 1 | 5 | 6
  IGF≥ 1.3 ULN | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Maintain Their Biochemical Response at the End of the Double Blind Placebo Controlled (DPC) Period.
Description: Maintenance of response was defined by using the average IGF-1 level of the last 2 available assessments in the DPC period. If the average IGF-1 is ≤ 1×ULN, a patient was classified as a responder (i.e., maintained their biochemical response). If the average IGF-1 is > 1×ULN, a patient was classified as a non-responder. Patients who discontinue study medication during the DPC period for any reason was classified as non-responders for the primary analysis, regardless of their IGF-1 values.
Time Frame: Week 36
Population: Number of Patients who Maintained Their Biochemical Response at the End of the DPC Period
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Capsules | Matching Placebo
Number analyzed (Participants) | 28 | 28
Participants | 16 | 5
Statistical Analysis 1: Comparison: Octreotide Capsules vs Matching Placebo; The proportion of [IGF-1/GH] responders was compared between treatment groups using an exact logistic regression model with categorical covariates for treatment group, prior SRL dose, and baseline [IGF-1/GH] level; Test type: Superiority; p = 0.0079, Regression, Logistic; The adjusted proportion of responders is 58.16 for Octreotide Capsule Treatment Group vs. 19.42 for the Placebo

2. Secondary Outcome: Number of Patients Who Maintain Growth Hormone (GH) Response at the End of the Double Blind Placebo Controlled Period
Description: Maintenance of GH response was defined as having mean Growth Hormone (5 measurements 30 minutes apart) < 2.5 ng/mL at the end of the double blind placebo controlled period, out of those who were responders on Somatostatin Receptor Ligands (SRLs) injections at Screening.
Time Frame: Week 36
Population: Number of patients who maintain Growth Hormone (GH) response at the end of the double blind placebo controlled period
Measure: Count of Participants; unit: Participants
Groups:
- Octreotide Capsules: Octreotide capsules 40mg/day, 60mg/day, 80 mg/day (individual dose titration)
- Placebo: Matching placebo
Arm/Group | Octreotide Capsules | Placebo
Number analyzed (Participants) | 28 | 28
Participants | 21 | 7
Statistical Analysis 1: Comparison: Octreotide Capsules vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0007, Regression, Logistic; The adjusted proportion of responders is 77.66 for Octreotide Capsule Treatment Group vs. 30.40 for the Placebo

3. Secondary Outcome: Number of Patients Who Begin Rescue Treatment
Description: Number of Patients who Began Rescue Treatment Prior to and Including Week 36
Time Frame: Week 36
Population: The number of patients who began rescue treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Octreotide Capsules | Placebo
Number analyzed (Participants) | 28 | 28
Participants | 7 | 19
Statistical Analysis 1: Comparison: Octreotide Capsules vs Placebo; Test type: Superiority; p = 0.0029, Fisher Exact

ADVERSE EVENTS:
Time Frame: 1 year, 10 months
Description: Safety population: All participants enrolled in the study who received any amount of the study drug.
Arm/Group | Octreotide Capsules | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/28
Serious Adverse Events (participants affected / at risk) | 2/28 | 1/28
Other Adverse Events (participants affected / at risk) | 28/28 | 27/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide Capsules (N=28) | Matching Placebo (N=28)
Cholecystitis acute (Hepatobiliary disorders) | 1 (2) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Octreotide Capsules (N=28) | Matching Placebo (N=28)
Abdominal discomfort (Gastrointestinal disorders) | 4 (4) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 2 (3) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 3 (3)
Constipation (Gastrointestinal disorders) | 3 (4) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 8 (9) | 6 (6)
Dyspepsia (Gastrointestinal disorders) | 3 (3) | 1 (2)
Flatulence (Gastrointestinal disorders) | 1 (1) | 2 (2)
Large intestinal polyp (Gastrointestinal disorders) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 6 (7) | 3 (3)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4) | 0 (0)
Fatigue (General disorders) | 2 (2) | 7 (8)
Influenza-like illness (General disorders) | 0 (0) | 2 (2)
Oedema peripheral (General disorders) | 2 (2) | 3 (3)
Pain (General disorders) | 2 (2) | 0 (0)
Peripheral swelling (General disorders) | 3 (4) | 4 (4)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1)
Nasopharyngitis (Infections and infestations) | 3 (3) | 4 (5)
Sinusitis (Infections and infestations) | 3 (3) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (6) | 1 (2)
Blood glucose increased (Investigations) | 3 (5) | 1 (2)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 3 (4)
Insulin-like growth factor increased (Investigations) | 0 (0) | 2 (2)
Weight increased (Investigations) | 2 (2) | 2 (2)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 (11) | 16 (28)
Arthritis (Musculoskeletal and connective tissue disorders) | 2 (3) | 2 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Soft tissue swelling (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Carpal tunnel syndrome (Nervous system disorders) | 4 (5) | 4 (5)
Headache (Nervous system disorders) | 4 (7) | 9 (17)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Paraesthesia (Nervous system disorders) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 1 (2) | 2 (2)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 (10) | 7 (8)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT03252353/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-29): https://cdn.clinicaltrials.gov/large-docs/53/NCT03252353/SAP_001.pdf